CLINICAL TRIAL: NCT04098978
Title: Before-after Comparison of Pharmacist Drug Therapy Management in Pediatric Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisiana Monroe (Other)
Collaborators: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hypertension; Blood Pressure
Keywords: Children; Adolescents; Young Adults; Pediatric Hypertension; Pharmacoeconomics; Pharmacist
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Before-after comparison of intervention to traditional care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist Drug Therapy Management (Experimental)
  Interventions: Other: Pharmacist Drug Therapy Management

INTERVENTIONS:
Other: Pharmacist Drug Therapy Management — Patients will be seen by pharmacist for collaborative drug therapy management.

SUMMARY:
This study will measure the effect of a novel pharmacy practice model on pediatric patients with hypertension. In North Louisiana, many patients have to travel to see subspecialists for treatment for hypertension and elevated blood pressure, which has many costs including direct medical costs, direct nonmedical costs, and indirect costs like missed time from work, school, or social obligations. Also, many patients who have to travel to get to their appointments have a high rate of missed appointments, which can be bad for overall health.

This study will use a pharmacist to perform collaborative drug therapy management with pediatric cardiologists to manage therapy for patients with hypertension or elevated blood pressure. Patients will monitor blood pressure at home and follow up with the pharmacist by telecommunications. Pharmacist drug therapy management and telemedicine have been studied separately, but this is the first study with pharmacist drug therapy management by telemedicine for pediatric patients. If this model is successful, it could be replicated in other rural areas to improve patient care and reduce healthcare costs.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of elevated blood pressure or hypertension.
* Physician decision to treat with drug therapy or lifestyle modifications and physician referral to pharmacist.
* Consent both to therapy with pharmacist and participation in study (Note: in the state of Louisiana, patients must provide consent to be treated in a collaborative drug therapy management program).
* For patients younger than 18, informed assent and parental permission to participate in the study. For patients who turn 18 during the study, informed consent will be obtained on the first visit after they turn 18.
* Males and females; age 4-20 at enrollment
* Willingness to adhere to study regimen

The same inclusion criteria will apply to control patients except that:

* They will have been treated at the clinic for hypertension or elevated blood pressure during the control period.
* A waiver of consent has been obtained for historical data.

Exclusion Criteria:

* Physical preclusion to taking blood pressure, such as lack of limbs or any congenital or acquired anatomical defect preventing routine measurement of blood pressure
* Participation in another treatment or intervention study for hypertension during the study period
* Inability to speak English
* For patients under 18 years old, not having at least one parent or guardian able to speak English
* Patients who are pregnant

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 266 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adequately-controlled hypertension at 3 months. | 3 months
Proportion of patients with adequately-controlled hypertension at 6 months. | 6 months
Proportion of patients with adequately-controlled hypertension at 12 months. | 12 months
Time to adequate control of hypertension. | Through study completion, an average of 1 year.
  Defined as the first appointment with controlled hypertension.

SECONDARY OUTCOMES:
Appointment adherence | Through study completion, an average of 1 year.
  Proportion of appointments attended
Number and type of serious adverse drug events | Through study completion, an average of 1 year.
  Number of serious adverse drug events in aggregate and subgrouped.
Number of unplanned health care encounters related to hypertension | Through study completion, an average of 1 year.
  Surrogate for adverse event associated with treatment or disease state.
Costs to patients | Through study completion, an average of 1 year.
  Includes direct medical, direct nonmedical, indirect costs
Costs to communities | Through study completion, an average of 1 year.
  Includes healthcare resource utilization, lost productivity
Cost to healthcare systems and payors | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Health Center for Children, West Monroe, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be available to researchers within the University of Louisiana Monroe based on IRB review and approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon completion of study.

REFERENCES:
- [Background] Syed ST, Gerber BS, Sharp LK. Traveling towards disease: transportation barriers to health care access. J Community Health. 2013 Oct;38(5):976-93. doi: 10.1007/s10900-013-9681-1. PMID 23543372
- [Background] Stumetz KS, Yi-Frazier JP, Mitrovich C, Briggs Early K. Quality of care in rural youth with type 1 diabetes: a cross-sectional pilot assessment. BMJ Open Diabetes Res Care. 2016 Nov 24;4(1):e000300. doi: 10.1136/bmjdrc-2016-000300. eCollection 2016. PMID 27933188
- [Background] Dalton K, Byrne S. Role of the pharmacist in reducing healthcare costs: current insights. Integr Pharm Res Pract. 2017 Jan 25;6:37-46. doi: 10.2147/IPRP.S108047. eCollection 2017. PMID 29354549
- [Background] Hawes EM, Misita C, Burkhart JI, McKnight L, Deyo ZM, Lee RA, Howard C, Eckel SF. Prescribing pharmacists in the ambulatory care setting: Experience at the University of North Carolina Medical Center. Am J Health Syst Pharm. 2016 Sep 15;73(18):1425-33. doi: 10.2146/ajhp150771. PMID 27605321
- [Background] Kruse CS, Krowski N, Rodriguez B, Tran L, Vela J, Brooks M. Telehealth and patient satisfaction: a systematic review and narrative analysis. BMJ Open. 2017 Aug 3;7(8):e016242. doi: 10.1136/bmjopen-2017-016242. PMID 28775188
- [Background] Victor RG, Lynch K, Li N, Blyler C, Muhammad E, Handler J, Brettler J, Rashid M, Hsu B, Foxx-Drew D, Moy N, Reid AE, Elashoff RM. A Cluster-Randomized Trial of Blood-Pressure Reduction in Black Barbershops. N Engl J Med. 2018 Apr 5;378(14):1291-1301. doi: 10.1056/NEJMoa1717250. Epub 2018 Mar 12. PMID 29527973
- [Background] Weeks G, George J, Maclure K, Stewart D. Non-medical prescribing versus medical prescribing for acute and chronic disease management in primary and secondary care. Cochrane Database Syst Rev. 2016 Nov 22;11(11):CD011227. doi: 10.1002/14651858.CD011227.pub2. PMID 27873322
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Flinn SK, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017 Sep;140(3):e20171904. doi: 10.1542/peds.2017-1904. Epub 2017 Aug 21. PMID 28827377
- [Background] Chen X, Wang Y. Tracking of blood pressure from childhood to adulthood: a systematic review and meta-regression analysis. Circulation. 2008 Jun 24;117(25):3171-80. doi: 10.1161/CIRCULATIONAHA.107.730366. Epub 2008 Jun 16. PMID 18559702
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, et al; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017; 140(3):e20171904. Pediatrics. 2017 Dec;140(6):e20173035. doi: 10.1542/peds.2017-3035. No abstract available. PMID 29192011
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] Twigg G, Motsko J, Thomas J, David T. Pharmacist-Managed Diabetes Center Interventions Ensure Quality and Safety in Elderly Patients. Consult Pharm. 2017 May 1;32(5):299-310. doi: 10.4140/TCP.n.2017.299. PMID 28483010